CLINICAL TRIAL: NCT05652140
Title: Cardiorespiratory Fitness and the Apolipoprotein E (ApoE) Genotype and Its Interaction With Cognitive Functions and Cognitive Decline in Late-Middle-Aged Older Adults: A Prospective Study
Brief Title: Cardiorespiratory Fitness, Apolipoprotein E Genotype, and Cognitive Functions: A Prospective Study
Status: Completed | Type: Observational
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yu-Kai Chang, Professor, National Taiwan Normal University
Other Study IDs: PACNL_APOE_PROSPECTIVE
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Aging; Cognitive Change
Keywords: physical fitness; Apolipoprotein E; event-related potential

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- High-Risk with increased CRF: ApoE e4 carriers with increased CRF from Baseline to the Follow-Up Stages.
  Interventions: Other: Data collections
- High-Risk with decreased CRF: ApoE e4 carriers with decreased CRF from Baseline to the Follow-Up Stages.
  Interventions: Other: Data collections
- Low-Risk with increased CRF: Non-ApoE e4 carriers with increased CRF from Baseline to the Follow-Up Stages.
  Interventions: Other: Data collections
- Low-Risk with decreased CRF: Non-ApoE e4 carriers with decreased CRF from Baseline to the Follow-Up Stages.
  Interventions: Other: Data collections

INTERVENTIONS:
Other: Data collections — Data collections of cognitive function, neuroelectrical activities, ApoE genotype, and physical fitness.

SUMMARY:
The current research project aims to investigate the interaction of cardiorespiratory fitness (CRF) and the ApoE genotype with neurocognitive functions.

DETAILED DESCRIPTION:
The current research project aims to investigate the interaction of cardiorespiratory fitness (CRF) and the ApoE genotype with neurocognitive functions. The three main purposes of the current research project seek to achieve:

1. An exploration of the associations of, as well as the interactions between, CRF assessed at the Baseline Stage, and the ApoE genotype, along with cognitive functions in cognitively healthy late-middle-aged older adults.
2. The employing of an event-related potential (ERP) to investigate the associations between the baseline CRF, the ApoE genotype, and cognitive functions in cognitively healthy late-middle-aged older adults, as well as the potential underlying neuroelectrical mechanisms.
3. An investigation of the interactions between the changes of CRFs assessed at the Baseline and the Follow-Up Stages and the ApoE genotype in relation to neurocognitive function, as well as the underlying neuroelectrical mechanisms, in cognitively healthy late-middle-aged older adults.

ELIGIBILITY:
Inclusion Criteria:

* right handed
* no history of cardiorespiratory disease
* normal or corrected-to-normal vision based on the 20/20 standard
* no risk of performing physical activities, as measured by the Physical Activity Readiness Questionnaire

Exclusion Criteria:

* the scores of Mini-Mental Status Examination (MMSE) < 25 and cognitively intact upon study entry
* history of psychiatric or neurological diseases
* color-blindness

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cognitively healthy late-middle-aged older adults recruited from the northern part of Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, Ph.D., Study Director — Department of Physical Education and Sport Sciences, National Taiwan Normal University
Locations (1):
- Department of Physical Education and Sport Sciences, National Taiwan Normal University, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-Risk With Decreased CRF | High-Risk With Increased CRF | Low-Risk With Decreased CRF | Low-Risk With Increased CRF
Started | 22 | 21 | 57 | 59
Completed | 15 | 5 | 35 | 28
Not Completed | 7 | 16 | 22 | 31
Not completed — Lost to Follow-up | 7 | 16 | 22 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Risk With Decreased CRF | High-Risk With Increased CRF | Low-Risk With Decreased CRF | Low-Risk With Increased CRF | Total
Number analyzed (Participants) | 22 | 21 | 57 | 59 | 159
Age, Customized [Number; unit: participants]
  Aged between 50-70 year-old | 22 | 21 | 57 | 59 | 159
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 44 | 45 | 120
  Male | 7 | 5 | 13 | 14 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 21 | 57 | 59 | 159
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 22 | 21 | 57 | 59 | 159
Stroop response time (RT) [Mean (Standard Deviation); unit: ms] — Response time (RT) during the incongruent trials was recorded as one of the behavioral indexes.
  ms | 730.68 (84.52) | 678.90 (86.19) | 722.12 (86.13) | 701.81 (67.91) | 710.06 (80.49)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Inhibitory Performance: Stroop Task
Description: Inhibitory performance was assessed using the computerized Stroop task at the Baseline and at the Follow-Up assessments. The difference in response time (RT) between the Baseline and the Follow-Up Stages was calculated as the index of the inhibitory performance.
Time Frame: 30 minutes each at the Baseline and the Follow-Up visit at Month 18
Measure: Mean (Standard Error); unit: ms
Arm/Group | High-Risk With Decreased CRF | High-Risk With Increased CRF | Low-Risk With Decreased CRF | Low-Risk With Increased CRF
Number analyzed (Participants) | 15 | 5 | 35 | 28
ms | 1.66 (13.30) | -29.85 (3.21) | 21.49 (8.75) | -20.13 (9.78)

2. Primary Outcome: Changes in Neuroelectrical Activities
Description: The neuroelectrical activities (P3 component) during the Stroop task were recorded and analyzed using the Neuroscan system. The difference in P3 amplitudes of incongruent trials between the Baseline and the Follow-Up Stages was calculated as the index of the neuroelectrical index.
Time Frame: 30 minutes each at the Baseline and the Follow-Up visit at Month 18
Measure: Mean (Standard Error); unit: microvolt
Arm/Group | High-Risk With Decreased CRF | High-Risk With Increased CRF | Low-Risk With Decreased CRF | Low-Risk With Increased CRF
Number analyzed (Participants) | 15 | 5 | 35 | 28
microvolt | -1.80 (0.90) | 2.81 (1.76) | -1.20 (0.61) | 0.57 (0.67)

3. Secondary Outcome: Number of Participants for Whom ApoE Genotype Was Determined
Description: Participants' ApoE genotype was determined based on the genetic biomarkers (rs429358 and rs7412)
Time Frame: 5 minutes at the Baseline Stage.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Risk With Decreased CRF | High-Risk With Increased CRF | Low-Risk With Decreased CRF | Low-Risk With Increased CRF
Number analyzed (Participants) | 22 | 21 | 57 | 59
Participants | 22 | 21 | 57 | 59

4. Secondary Outcome: Physical Fitness Measurements: Changes in Aerobic Fitness
Description: Participants' aerobic fitness was estimated using the submaximal cycle ergometer test at the baseline and at the follow-up assessments. The difference in maximum oxygen consumption (VO2 max) between the Baseline and the Follow-Up Stages was calculated as the index of aerobic fitness.
Time Frame: 30 minutes each at the Baseline and the Follow-Up visit at Month 18
Measure: Mean (Standard Error); unit: ml·kg-1·min-1
Arm/Group | High-Risk With Decreased CRF | High-Risk With Increased CRF | Low-Risk With Decreased CRF | Low-Risk With Increased CRF
Number analyzed (Participants) | 15 | 5 | 35 | 28
ml·kg-1·min-1 | -4.03 (3.18) | 1.52 (2.08) | -4.76 (3.65) | 3.28 (4.29)

5. Other Pre Specified Outcome: Changes in Higher Order Executive Performance: Tower of London Test
Description: Higher order executive performance was assessed using the Tower of London Test at the baseline and at the follow-up assessments. Changes in higher order executive performance from Baseline to the Follow-Up Stages were assessed.
Time Frame: 30 minutes each at the Baseline and the Follow-Up Stages.
Population: The Tower of London Test, a pre-specified Primary Outcome Measure, was not administered to any participants due to unforeseen constraints in practical resource availability at the study sites (i.e., unavailability of required test materials and time limitations that precluded its inclusion within the study timeline). Consequently, no data was collected for this outcome measure.
Arm/Group | High-Risk With Decreased CRF | High-Risk With Increased CRF | Low-Risk With Decreased CRF | Low-Risk With Increased CRF
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2.5 years.
Arm/Group | High-Risk With Increased CRF | High-Risk With Decreased CRF | Low-Risk With Increased CRF | Low-Risk With Decreased CRF
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/57 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/57 | 0/59
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/57 | 0/59

LIMITATIONS AND CAVEATS:
Due to the substantial overlapping of the study period with the COVID-19 pandemic, a larger-than-expected number of participants withdrew following the completion of the baseline stage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT05652140/Prot_SAP_000.pdf